CLINICAL TRIAL: NCT03598244
Title: A Phase I Study of Savolitinib in Recurrent, Progressive or Refractory Medulloblastoma, High-Grade Glioma, Diffuse Intrinsic Pontine Glioma, and CNS Tumors Harboring MET Aberrations
Brief Title: Volitinib in Treating Patients With Recurrent or Refractory Primary CNS Tumors
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2018-01499; NCI-2018-01499 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); PBTC-049 (Other: Pediatric Brain Tumor Consortium); PBTC-049 (Other: CTEP); UM1CA081457 (NIH)
Record Dates: First submitted 2018-07-24; First posted 2018-07-26 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Recurrent Diffuse Intrinsic Pontine Glioma; Recurrent Malignant Glioma; Recurrent Medulloblastoma; Recurrent Primary Central Nervous System Neoplasm; Refractory Diffuse Intrinsic Pontine Glioma; Refractory Malignant Glioma; Refractory Medulloblastoma; Refractory Primary Central Nervous System Neoplasm
MeSH Terms: conditions — Diffuse Intrinsic Pontine Glioma; Glioma; Medulloblastoma; Central Nervous System Neoplasms | interventions — Specimen Handling; Magnetic Resonance Spectroscopy; 1-(1-(imidazo(1,2-a)pyridin-6-yl)ethyl)-6-(1-methyl-1H-pyrazol-4-yl)-1H-(1,2,3)triazolo(4,5-b)pyrazine; X-Rays; Phantoms, Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (volitinib) (Experimental): Patients receive volitinib PO QD. Treatment repeats every 28 days for up to 39 courses in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo blood sample collection, X-ray imaging, and MRI scans throughout study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Magnetic Resonance Imaging; Drug: Savolitinib; Procedure: X-Ray Imaging

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Magnetic Resonance Imaging — Undergo MRI scan
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Drug: Savolitinib — Given PO
  Other Names: AZD 6094; AZD6094; HMPL-504; Volitinib
Procedure: X-Ray Imaging — Undergo X-ray imaging
  Other Names: Conventional X-Ray; Diagnostic Radiology; Medical Imaging, X-Ray; Plain film radiographs; Radiographic Imaging; Radiographic imaging procedure (procedure); Radiography; RG; Static X-Ray; X-Ray

SUMMARY:
This phase I trial studies the side effects and best dose of volitinib in treating patients with primary central nervous system (CNS) tumors that have come back (recurrent) or does not respond to treatment (refractory). Volitinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate the maximum tolerated dose (MTD) and recommend a phase II dose of volitinib (savolitinib) administered orally daily in children with refractory, progressive or recurrent primary CNS tumors.

II. To define and describe the toxicities of savolitinib in children with refractory, progressive, or recurrent primary CNS tumors.

III. To characterize the pharmacokinetics of savolitinib in children with refractory, progressive, or recurrent primary CNS tumors.

SECONDARY OBJECTIVES:

I. To preliminarily define the antitumor activity of savolitinib within the confines of a phase I study.

II. To perform a genomic analysis within the confines of a phase I study to investigate correlation between response to treatment (as measured by objective response or progression free survival [PFS]) and the presence of specific genomic alterations (e.g., MET or HGF amplification, MET mutations, or MET fusion) and/or specific subgroups of disease.

OUTLINE: This is a dose-escalation study of volitinib followed by a dose-expansion study.

Patients receive volitinib orally (PO) once daily (QD). Treatment repeats every 28 days for up to 39 courses in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo blood sample collection X-ray imaging, and magnetic resonance imaging (MRI) scans throughout study.

After completion of study treatment, patients are followed up at 30 days, then periodically for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a histologically confirmed diagnosis of a primary CNS tumor (medulloblastoma, high-grade glioma, or diffuse intrinsic pontine glioma [DIPG]) that is recurrent, refractory, or progressive. All tumors must have histologic verification at either the time of diagnosis or recurrence except patients with diffuse intrinsic brain stem tumors. These patients must have radiographic or clinical evidence of progression. Patients with a recurrent, progressive, or refractory primary CNS tumor with evidence of genetic activation of the MET pathway, regardless of histology, are also eligible to the Phase I component of this study

  * Note: Refractory disease is defined as the presence of persistent abnormality on conventional MRI imaging that is further distinguished by histology (biopsy or sample of lesion) or advanced imaging, OR as determined by the treating physician and discussed with the primary investigator prior to enrollment
* Efficacy Expansion Cohort: Patients must have a recurrent, progressive, or refractory primary CNS tumor with evidence of genetic activation of the MET pathway, regardless of histology. Specimens can be from diagnosis or recurrence and there is no time limit from when the specimen was obtained prior to enrollment onto the efficacy expansion cohort. Results from a Clinical Laboratory Improvement Act (CLIA)-certified laboratory will be accepted for this eligibility criterion. Sites must provide a redacted copy of the local CLIA-certified sequencing laboratory report to the study chair via email prior to enrollment. MET pathway activation is defined as:

  * MET mutations, OR
  * MET or HGF amplification, OR
  * MET fusion
* Recurrent or refractory primary malignant CNS tumor patients must have adequate pre-trial frozen or formalin-fixed paraffin-embedded (FFPE) tumor material available for the required correlative studies. If target amounts of tissue or number of slides are not available, the site must obtain study chair/co-chair approval for adequacy of submitted tumor samples and prioritization of studies to be performed, prior to patient enrollment

  * Patients with DIPG who have pre-trial tumor tissue available are requested to submit tissue; however, this is not required for eligibility
* Patients must have evaluable disease to be eligible. Evaluable disease is defined as the presence of at least one lesion that can be measured accurately in at least 2 (two) dimensions
* Patients must be > 5 years and =< 21 years of age at the time of study enrollment
* Body surface area (BSA)

  * Patients enrolled on 75 mg/m^2/day (dose level 0) must have a BSA >= 1.00 m^2
  * Patients enrolled on 150 mg/m^2/day (dose level 1) must have a BSA >= 0.55 m^2
  * Patients enrolled on 240 mg/m^2/day (dose level 2) must have a BSA >= 0.67 m^2
  * Patients enrolled on 350 mg/m^2/day (dose level 3) must have a BSA >= 0.73 m^2
* Patients must have failed prior standard therapy for their tumor. Patients with medulloblastoma must have received radiation therapy in addition to platinum and alkylator-based chemotherapy. Patients with high-grade glioma (HGG) and DIPG must have at least received radiation therapy. Patients must have recovered from the acute treatment related toxicities (defined as =< grade 1 if not defined in eligibility criteria) of all prior chemotherapy, immunotherapy, radiotherapy, or any other treatment modality prior to entering this study
* Patients must have received their last dose of known myelosuppressive anticancer therapy at least 21 days prior to enrollment or at least 42 days if it included nitrosourea
* Biologic or investigational agent (anti-neoplastic):

  * Patients must have recovered from any acute toxicity potentially related to the agent and received their last dose of the investigational or biologic agent >= 7 days prior to study enrollment

    * For agents that have known adverse events occurring beyond 7 days after administration, this period must be extended beyond the time during which adverse events are known to occur

Monoclonal antibody treatment and agents with known prolonged half-lives:

* Patients must have recovered from any acute toxicity potentially related to the agent and received their last dose of the agent >= 28 days prior to study enrollment

  * Patients must have had their last fraction of:
* Craniospinal irradiation or total body irradiation or radiation to >= 50% of pelvis > 12 weeks prior to enrollment
* Focal irradiation > 4 weeks prior to enrollment

  * Patients must be:
* >= 24 weeks since allogeneic stem cell transplant prior to enrollment with no evidence of active graft versus (vs.) host disease
* >= 12 weeks since autologous stem cell transplant prior to enrollment

  * Neurologic Status
* Patients with neurological deficits should have deficits that are stable for a minimum of 1 week prior to enrollment. A baseline detailed neurological exam should clearly document the neurological status of the patient at the time of enrollment on the study
* Patients with seizure disorders may be enrolled if seizures are well controlled
* Patients must be able to swallow whole tablets to be eligible for study enrollment

  * Karnofsky performance scale (KPS for > 16 years of age) or Lansky performance score (LPS for =< 16 years of age) assessed within two weeks of enrollment must be >= 50
* Patients who are unable to walk because of neurologic deficits, but who are up in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score

  * Absolute neutrophil count >= 1.0 x 10^9 cells/ L
  * Platelets >= 100 x 10^9 cells/ L (unsupported, defined as no platelet transfusion within 7 days prior to enrollment)
  * Hemoglobin >= 8 g/dL (hemoglobin should be unsupported, i.e., red blood cell transfusions are not allowed within 14 days prior to enrollment)
  * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) =< 2.5 x the upper limit of normal (ULN) with total bilirubin =< 1x ULN OR total bilirubin > ULN - =< 1.5 x ULN with ALT and AST =< 1 x ULN
  * Albumin >= 2 g/dL
  * Serum creatinine based on age/gender. Patients that do not meet the criteria below but have a 24 hour creatinine clearance or glomerular filtration rate (GFR) (radioisotope or iothalamate) >= 70 mL/min/1.73 m^2 are eligible
* Age: Maximum serum creatinine (mg/dL)
* 2 to < 6 years: 0.8 (male and female)
* 6 to < 10 years: 1 (male and female)
* 10 to < 13 years: 1.2 (male and female)
* 13 to < 16 years: 1.5 (male), 1.4 (female)
* >= 16 years: 1.7 (male), 1.4 (female)

  * International normalized ratio (INR) < 1.5 x ULN and activated partial thromboplastin time (aPTT) < 1.5 x ULN unless patients are receiving therapeutic anti-coagulation which affects these parameters
  * Patients with known tumor thrombus or deep vein thrombosis are eligible if clinically stable on low molecular weight heparin for >= 2 weeks
  * Cardiac function:
* Mean resting corrected QT interval (QTc Bazett) =< 450 msec on screening obtained from 3 electrocardiograms (EKGs)

  * Oxygen saturation as measured by pulse oximetry is > 93% on room air
  * Patients who are receiving corticosteroids must be on a stable or decreasing dose for at least 1 week prior to enrollment
  * Patients must be off all colony-stimulating factor(s) (e.g., filgrastim, sargramostim or erythropoietin) for at least 1 week prior to enrollment. Two (2) weeks must have elapsed if patients received polyethylene glycol (PEG) formulations
  * Pregnancy Prevention
* Patients of childbearing or child fathering potential must be willing to use a medically acceptable form of birth control, which includes abstinence, while being treated on this study
* Women of child-bearing potential should use effective contraception from the time of enrollment until 4 weeks after discontinuing study treatment
* Male study participants should use a condom with female partners of child-bearing potential during the study and for 24 weeks after discontinuing study treatment
* If the female partner of a male study participant is not using effective contraception, men must use a condom during the study and for 24 weeks after discontinuing study treatment
* Male study participants should avoid fathering a child and refrain from sperm donation from study start to 24 weeks after discontinuing study treatment

  * Ability to understand and willingness to sign a written informed consent document. Legally authorized representatives may sign and give informed consent on behalf of study participants

Exclusion Criteria:

* Pregnant women or nursing mothers are excluded from this study. Female patients of childbearing potential must have a negative serum or urine pregnancy test within 7 days prior to enrollment. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required. Pregnant women are excluded from this study because there are unknown but potential risks to an unborn baby from savolitinib. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with savolitinib, breastfeeding should be discontinued if the mother is treated with savolitinib
* Patients with a known serious active infection including, but not limited to human immunodeficiency virus, and tuberculosis
* Patients with a known active or resolved viral hepatitis infection
* Patients with any clinically significant unrelated systemic illness or significant cardiac, pulmonary, hepatic, or other organ dysfunction), that in the opinion of the investigator would compromise the patient's ability to tolerate protocol therapy, put them at additional risk for toxicity or would interfere with the study procedures or results
* Patients with uncontrolled hypertension (i.e., a blood pressure [BP] > 95th percentile for age, height, and gender, patients with values above these levels must have their blood pressure controlled with medication prior to starting study drug)

  * The normal blood pressure by height, age, and gender can be assessed by using the NIH Guidelines on the PBTC Member's website (Protocols- Generic Forms and Templates- Normal Blood Pressure by Height and Age)
* Patients with any of the following cardiac diseases

  * Congestive heart failure (New York Heart Association >= grade 2)
  * Clinically significant cardiac arrhythmia
  * Mean resting corrected QT interval (QTc Bazett) > 450 msec on screening obtained from 3 electrocardiograms (EKGs) or
  * Factors that may increase the risk of QTc prolongation such as chronic hypokalemia not correctable with supplements, congenital or familial long QT syndrome, or
  * Family history of unexplained sudden death under 40 years of age in first-degree relatives or
  * Any concomitant medication known to prolong the QT interval and cause Torsade de Pointes. These drugs must have been discontinued prior to the start of administration of study treatment in accordance with guidance
  * Any clinically important abnormalities in rhythm, conduction, or morphology of resting EKG, e.g., complete left bundle branch block, third degree heart block, second degree heart block, PR interval > 250 msec
* Patients with history of liver cirrhosis of any origin and clinical stage; or history of other serious liver disease or chronic disease with relevant liver involvement, with or without normal liver function tests (LFTs), including but not limited to:

  * Hemochromatosis
  * Alpha -1 antitrypsin deficiency
  * Autoimmune hepatitis (AIH)
  * Primary sclerosing cholangitis (PSC)
  * Primary biliary cirrhosis (PBC)
  * Biopsy-confirmed non-alcoholic steatohepatitis (NASH) with advanced fibrosis
  * Biopsy-confirmed alcoholic steatohepatitis with advanced fibrosis
  * Wilson's disease
  * Hepatocellular carcinoma

    * Patients with liver metastases are eligible, provided they meet other eligibility criteria, including liver biochemistry criteria
* Patients with a prior or concurrent malignancy whose natural history or treatment has the potential to interfere with the safety or efficacy assessment of the investigational regimen for this trial
* Concurrent Therapy

  * Patients who are receiving any other anticancer or investigational drug therapy
  * Patients receiving strong inducers of CYP3A4, strong inhibitors of CYP3A4 or CYP1A2 or CYP3A4 substrates with a narrow therapeutic index within 2 weeks of the first dose of savolitinib (3 weeks for St John's Wort). Strong inducers of CYP3A4 and CYP3A4 substrates which have a narrow therapeutic range or CYP3A4 sensitive substrates should not be used during the trial or used with caution. Because the lists of these agents are constantly changing, it is important to regularly consult a frequently-updated medical reference. Patient drug information handout and wallet card should be provided to patients
  * Prior or current treatment with a MET inhibitor (e.g., foretinib, crizotinib, cabozantinib, or onartuzumab)
* Patient is currently receiving any of the following herbal preparations or medications and cannot be discontinued 1 week (7 days) prior to enrollment (3 weeks for St. John's wort). These herbal medications include, but are not limited to: cannabis products, St. John's wort, kava, ephedra (ma huang), gingko biloba, dehydroepiandrosterone (DHEA), yohimbe, saw palmetto, and ginseng
* Patient has undergone major surgical procedure =< 28 days prior to beginning study drug or a minor surgical procedure =< 7 days prior to beginning study drug. No waiting is required following port-a-cath placement
* Patients who in the opinion of the investigator are unwilling or unable to return for required follow-up visits or obtain follow-up studies required to assess toxicity to therapy or to adhere to drug administration plan, other study procedures, and study restrictions
* Patients with a history of allergic reactions attributed to compounds of similar chemical or biologic composition
* Prisoners will be excluded from this study

Ages: 6 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 41 (Actual)
Dates: Start 2018-11-27 (Actual); Primary Completion 2025-04-14 (Actual); Study Completion 2026-04-14 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose of volitinib | Up to 30 days post treatment
  Will be defined as the highest dose level at which six patients have been treated with at most one patient experiencing a dose limiting toxicity and the next higher dose level has been determined to be too toxic.
Recommend phase II dose | Up to 30 days post treatment

SECONDARY OUTCOMES:
Objective responses (complete response + partial response) | Up to 2 years
  Will be described by dose and by histology. Prolonged stable diseases will also be reported in a descriptive fashion.
Molecular analyses of tumors | Up to 2 years
  Will be reported descriptively.
Pharmacokinetic Parameters | Up to 2 years
  Will be presented in tabular and graphical form. Pharmacokinetic parameters of interest, such as apparent volume of the central compartment (Vc/F), elimination rate constant (Ke), half-life (t1/2), apparent oral clearance (CL/F), and area under the plasma concentration time curve (AUC) will be estimated using compartmental methods. Dose proportionality in pharmacokinetic parameters will be investigated by performing one-way analysis of variance (ANOVA) on dose-normalized parameters.
Population parameters | Up to 2 years
  Will be estimated using nonlinear mixed effects modeling methods (NONMEM). This method estimates the population parameters and both the inter- and intra-subject variability. Once the population parameters and corresponding covariance matrix are estimated, individual estimates can be obtained using post hoc analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Ralph Salloum, Principal Investigator — Pediatric Brain Tumor Consortium
Locations (12):
- United States (11):
  - Children's Hospital Los Angeles, Los Angeles, California
  - Lucile Packard Children's Hospital Stanford University, Palo Alto, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Lurie Children's Hospital-Chicago, Chicago, Illinois
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Saint Jude Children's Research Hospital, Memphis, Tennessee
  - Texas Children's Hospital, Houston, Texas
- Hospital for Sick Children, Toronto, Ontario, Canada